CLINICAL TRIAL: NCT05082480
Title: A Prospective, Double-Centre, Randomized, Evaluator/Subject-blinded, Control Clinical Study: to Evaluate the Effectiveness of the Use of a Novel Crosslinking Hyaluronan Hydrogel on the Prevention of the Adhesion Occurrence After Trigger Finger Release Surgery
Brief Title: Evaluate the Effectiveness of Crosslinked HA on the Adhesion Preventing After Trigger Finger Release Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment
Sponsor: SciVision Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RDCT-TWDH
Record Dates: First submitted 2021-10-05; First posted 2021-10-19 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2022-05

CONDITIONS: Trigger Finger; Hyaluronic Acid
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic acid (HA) (Experimental): Hyaluronic acid (HA)
  Interventions: Device: Hyaluronic acid (HA)
- Saline (Placebo Comparator): Saline
  Interventions: Device: Saline

INTERVENTIONS:
Device: Hyaluronic acid (HA) — Hyaluronic acid (HA)
  Arms: Hyaluronic acid (HA)
Device: Saline — Saline
  Arms: Saline

SUMMARY:
To Evaluate the Effectiveness of the use of a Novel Crosslinking Hyaluronan Hydrogel on the Prevention of the Adhesion Occurrence After Trigger Finger Release Surgery

DETAILED DESCRIPTION:
The medical device is a bioabsorbable, extensible, crosslinked, 6% hyaluronic acid gel using fermentation sourced hyaluronic acid as a major component. This product could perfectly attach to the tissue surface, creating anti-adhesion layer which avoids post-surgical adhesion and is completely resorbed over time. This study is aimed to evaluate the effectiveness of the use of a novel crosslinking hyaluronan hydrogel on the prevention of the adhesion occurrence after trigger finger release surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to participate in this study and sign informed consent form
2. Age 20 to 65 years of male or female
3. The trigger finger, except thumb, classified as 3 to 4 points and plan to conduct trigger finger release surgery;
4. The trigger finger, except thumb, classified as 2 points with the symptom of flexion contracture and plan to conduct trigger finger release surgery;
5. Agree to comply with the follow-up schedule of this study

Exclusion Criteria:

1. Target finger has other adhesion in tendon, joint, or proximal nerve, neuropathy, compression injury or other disease;
2. Other fingers in the same hand as the target finger have other adhesion in tendon, joint, or proximal nerve, neuropathy, or compression injury;
3. Contralateral finger has other adhesion in tendon, joint, or proximal nerve, neuropathy, or compression injury;
4. The operation site was conducted tendon transplantation or any surgery in past 6 months;
5. Receiving orthopedic-related treatment which may affect the evaluation of the study;
6. The skin of the operation site with infection, deficiency, or needing skin transplantation;
7. With poorly controlled chronic diseases, such as diabetes mellitus;
8. Patient with autoimmune disease (such as rheumatoid arthritis), malignant tumors, coagulation diseases, heart diseases, mental diseases, etc., may cause patients to participate in the trial at higher risk;
9. Patient who has taken cortisol within the past 6 months, systemic corticosteroids within the past 2 months, immunosuppressive drugs within past 3 months, or non-steroidal anti-inflammatory drugs (NSAIDs) everyday within 1 week or NSAIDs within 8 hours occasionally. (subjects who have received inhaled/intranasal corticosteroids could be considered to include.);
10. With clinical meaningful coagulation disorders, underdoing anticoagulant treatment or taking blood circulation promotion and blood stasis removement medications within the past 10 days;
11. With history of hypersensitivity or allergy to hyaluronic acid or any component of the device; With history of hypersensitivity or allergy to Gram-positive bacteria or Streptococcus proteins; other severe hypersensitivity history unsuitable for participating in the study;
12. Pregnant, planning pregnancy or in breastfeeding females;
13. Other circumstances which judged to be unsuitable for participating in the study by the investigator.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
The percentage of Total Active Motion (TAM) score for target finger. | 30 days post-operation
  The percentage of Total Active Motion (TAM) score for target finger at 30 days post-operation.

SECONDARY OUTCOMES:
The percentage of TAM score of target finger. | baseline, 14, 60, 90, and 180 days post-operation
  The percentage of TAM score of target finger at baseline, 14, 60, 90, and 180 days post-operation.
TAM score of target finger. | baseline, 14, 30, 60, 90, and 180 days post-operation
  TAM score of target finger at baseline, 14, 30, 60, 90, and 180 days post-operation.
The grade of TAM score of target finger and contralateral finger. | baseline, 14, 30, 60, 90, and 180 days post-operation
  The grade of TAM score of target finger and contralateral finger at baseline, 14, 30, 60, 90, and 180 days post-operation
Subjects self-evaluating Visual Analogue Scale (VAS) in pain of target finger at baseline, 14, 30, 60, 90, and 180 days post-operation. | baseline, 14, 30, 60, 90, and 180 days post-operation
  Subjects self-evaluating Visual Analogue Scale (VAS) in pain of target finger at baseline, 14, 30, 60, 90, and 180 days post-operation. The VAS scale uses a 100 mm line labelled at '0' with 'no pain' and '100' with 'worst pain'
Subjects self-evaluating Quick Disabilities of the Arm, Shoulder and Hand Score (Quick-Dash). | baseline, 14, 30, 60, 90, and 180 days post-operation
  Subjects self-evaluating Quick Disabilities of the Arm, Shoulder and Hand Score (Quick-Dash) at baseline, 14, 30, 60, 90, and 180 days post-operation.
The evaluation of tendon by sonography. | baseline, 14, 30, 60, 90, and 180 days post-operation
  The evaluation of tendon by sonography at baseline, 14, 30, 60, 90, and 180 days post-operation.
Subjects self-evaluating Visual Analogue Scale (VAS) in satisfaction | 14, 30, 60, 90, and 180 days post-operation
  Subjects self-evaluating satisfaction at 14, 30, 60, 90, and 180 days post-operation. Patients rate their treatment satisfaction based on a 100 mm VAS. The VAS scale uses a 100 mm line labelled at '0' with 'least satisfaction' and '100' with 'highest satisfaction'.
The incidence, severity and correlation of adverse event (AE) and serious adverse event (SAE). | baseline, 14, 30, 60, 90, and 180 days post-operation
  The incidence, severity and correlation of adverse event (AE) and serious adverse event (SAE).

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Municipal Ta-Tung Hospital, Kaohsiung City

IPD SHARING:
Plan to Share IPD: No